CLINICAL TRIAL: NCT06621615
Title: An Open Label, Multicenter Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics, and Efficacy of CVL006 Injection in Patients With Advanced Solid Tumors.
Brief Title: Clinical Study of CVL006 Injection in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL006-T1001
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor
Keywords: Late stage solid tumor; DLT; MTD; RP2D

STUDY DESIGN:
Intervention Model Description: This study is a phase I clinical trial of dose escalation/dose extension/efficacy extension of CVL006 injection monotherapy in patients with advanced solid tumors in a single arm, open label, multicenter manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVL006 monotherapy group (Experimental): This study is divided into three stages. Ia. Dose escalation stage: Accelerated titration combined with a "3+3" design was used for dose escalation, with a maximum enrollment of 42 subjects.
  Ib. Dose extension stage: Based on the data from dose escalation, in dose groups where a certain therapeutic effect is observed, each dose group will be extended by no more than 10 subjects, and RP2D will be determined based on the data from dose escalation and extension stages.
  Ic. Efficacy expansion stage: RP2D was selected for expansion, with each tumor type expanded to 10-30 cases.
  The above three stages involve intravenous infusion of CVL006, administered every 2 weeks and every 28 days as a treatment cycle. The first treatment cycle (28 days) serves as the DLT observation period, during which DLT is collected and its MTD and RP2D are determined.
  Interventions: Biological: CVL006 Injection

INTERVENTIONS:
Biological: CVL006 Injection — CVL006 injection, intravenous infusion, administered every 2 weeks. Every 28 days is a cycle. Until the subject cannot tolerate the disease progression or toxicity, or the researcher determines that the medication must be terminated or the sponsor terminates the study. SMC can adjust the dosing frequency based on safety, tolerability, and PK results data. If researchers consider that subjects enrolled in the lower dose group can benefit from the study intervention, they can allow them to continue treatment at a higher dose that has been proven safe based on the researcher's judgment.
  Other Names: B006

SUMMARY:
Evaluate the safety and tolerability of CVL006 monotherapy in patients with advanced solid tumors; Observe the dose limiting toxicity (DLT) of CVL006 monotherapy in patients with advanced solid tumors, evaluate the maximum tolerated dose (MTD), and recommend the dosage for phase II clinical trials (RP2D).

DETAILED DESCRIPTION:
This study is a phase I clinical trial of single arm, open label, multicenter dose escalation/dose extension/efficacy extension. The research process for each dose group includes a screening period (from the signing of the informed consent form by the subjects to 1 day before the first study medication), a medication period (from the first study medication to termination of medication), and a follow-up period (90 days after termination of medication). This study is divided into three stages: I. Dose escalation stage: Accelerated titration combined with a "3+3" design is used to dose up CVL006 injection. Accelerated titration is preset with three doses, starting at 0.03 mg/kg. Only one subject is enrolled in each dose group. After completing the three preset doses, four dose groups are designed according to the "3+3" principle, with 3-6 subjects enrolled in each dose group, up to a maximum of 42 subjects enrolled. Ib. Dose extension stage: Based on the observed safety, tolerability, efficacy, and PK characteristics during the dose escalation process, in the dose group where a certain therapeutic effect is observed in the subjects (such as 1 PR/CR or 2 SD), the SMC meeting will decide whether to extend the dose in that dose group. Plan to expand each dose group by no more than 10 subjects (including subjects with the same dose during the dose escalation phase). And determine RP2D based on data from dose escalation and expansion stages. Ic. Efficacy expansion stage: RP2D was selected for expansion, with each tumor type expanded to 10-30 cases. This study is expected to enroll approximately 100-120 cases, depending on the actual situation. Dose escalation, dose expansion, and efficacy expansion are the same: CVL006 injection, intravenous infusion, once every 2 weeks, every 28 days as a cycle. The subsequent administration time is calculated based on the actual date of the previous CVL006 administration. SMC can adjust the dosing frequency based on safety, tolerability, and PK results data.

ELIGIBILITY:
Inclusion Criteria:

- Participants must meet all of the following inclusion criteria in order to be enrolled in this study

1. Age: 18~75 years old (including both ends), gender not limited;
2. Dose escalation and dose expansion stage: For patients with advanced malignant solid tumors confirmed by histology or cytology, if standard treatment has failed, or if there is no standard treatment plan, or if standard treatment is not applicable at this stage;

   Efficacy expansion stage: Requirements for different types of tumors are as follows:

   Queue 1: Non small cell lung cancer (NSCLC) Locally advanced, recurrent, or metastatic NSCLC confirmed by histology or cytology, except for subjects known to have other driver genes (including sensitive EGFR mutations, ALK fusion, ROS1 fusion, BRAF V600E mutations, NTRK fusion, RET fusion, etc.); The subject received platinum based treatment on the first line, but did not receive PD-1/PD-L1 inhibitor treatment and had previous treatment failures; Or it may be determined by researchers that first-line platinum based dual therapy is intolerant, but PD-L1 TPS is ≥ 1%; Queue 2: Malignant Solid Tumors of MSI-H/dMMR Subjects with locally advanced, recurrent, or metastatic MSI-H/dMMR malignant solid tumors confirmed by histology or cytology, such as colorectal cancer, head and neck squamous cell carcinoma, etc., will be discussed and determined by the researchers and sponsors based on safety, PK, and efficacy results.

   Queue 3: Based on previous data, determine the tumor type with good therapeutic effect or recommended by the researcher (such as TMB-H) Subjects with locally advanced, recurrent, or metastatic TMB-H malignant solid tumors confirmed by histology or cytology as inoperable will be discussed and determined by the researchers and the sponsor based on safety, PK, and efficacy results.
3. All subjects are required to provide tumor tissue samples for PD-L1 testing: tumor tissue samples should preferably be newly obtained. For subjects who cannot provide newly obtained tissue, they can provide tumor tissue samples archived within 3 years before the first study treatment. The sample type should be neutral formalin fixed, paraffin embedded [FFPE] tissue blocks or at least 6 unstained tumor tissue sections; If there are less than 6 pieces, it is necessary to consult with the sponsor and obtain their agreement before being allowed to be included in the group;
4. ECOG performance status (PS) score 0-1 points;
5. Predicted survival period ≥ 3 months
6. According to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1), having at least one measurable lesion;
7. Having sufficient bone marrow and organ function (without using any blood components and/or cell growth factors within 14 days prior to starting the study treatment):

   Hemoglobin (HB) ≥ 90 g/L; Neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 90 × 109/L； Total bilirubin<1.5×ULN (for subjects diagnosed with Gilbert syndrome, total bilirubin≤3×ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN (in patients with liver metastases, ALT and/or AST ≤5×ULN)； International normalized ratio (INR) and activated partial thromboplastin (APTT) time≤1.5×ULN; Qualitative analysis of urinary protein≤1+; Or urine protein qualitative≥2+, requiring 24-hour urine protein<1g
8. Women with fertility must agree to abstain from sexual activity (avoid heterosexual intercourse) or use effective contraception methods for at least 6 months from the time of signing the informed consent form until the last administration of the study drug. And within 7 days before starting the study treatment, the blood HCG test must be negative and must be non lactating (if the serum pregnancy test is positive, pregnancy must be ruled out and confirmed with the sponsor before inclusion);
9. For male patients whose partners are women of childbearing age, they must agree to abstain from sexual activity for at least 6 months from the signing of the informed consent form until the last administration of the study drug, or to use effective contraception methods. Male patients must also agree not to donate sperm during the same time period;
10. The patient voluntarily joined this study, signed an informed consent form, and showed good compliance.

Exclusion Criteria:

-

Subjects with any of the following conditions will not be included in this study:

1. Accompanied by untreated or active central nervous system (CNS) tumor metastasis. Subjects with a history of meningeal metastasis or current meningeal metastasis.

   -For CNS metastatic subjects, if the CNS tumor has received sufficient local treatment (surgery or radiotherapy); From the end of local treatment to the screening period, no progress was found on imaging examinations; The neurological symptoms of the subjects can be stable for at least 2 weeks before the first medication and do not require glucocorticoid treatment; You can participate in the research;
2. Patients with other malignant tumors within the five years prior to the first use of the investigational drug, except for fully treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, and papillary thyroid carcinoma after radical surgery;
3. If the researcher determines that the tumor lesion has a tendency to bleed, and the screening imaging examination shows that the subject has imaging evidence of tumor invasion or wrapping around large blood vessels;
4. Subjects who have previously used VEGF/PD-1 (PD-L1) bispecific antibodies;
5. Have serious cardiovascular and cerebrovascular diseases, including but not limited to:

   1. Severe cardiac rhythm or conduction abnormalities within 6 months prior to the first use of the investigational drug, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc;
   2. Within 6 months prior to the first use of the investigational drug, acute coronary syndrome, congestive heart failure (NYHA functional class ≥ II), and aortic dissection occurred;
   3. Within the first 6 months prior to the use of the investigational drug, there have been incidents of arteriovenous thrombosis, such as cerebrovascular accidents (transient ischemic attack, cerebral hemorrhage, stroke), deep vein thrombosis, and pulmonary embolism;
   4. Left ventricular ejection fraction (LVEF)<50% within 28 days prior to the first use of the investigational drug;
   5. In a resting state, the mean QTcF obtained from three baseline 12 (or more) lead electrocardiograms is greater than 470 ms for females or greater than 450 ms for males;
6. There is uncontrollable pleural effusion, abdominal effusion, or pericardial effusion;
7. Patients known or suspected to have interstitial pneumonia; Within three months prior to the first administration, other severe lung diseases that severely affect respiratory function, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/bronchiolitis obliterans; Non infectious pulmonary inflammation currently requiring steroid treatment;
8. Patients who have received immunotherapy in the past and have experienced ≥ grade 3 irAE or ≥ grade 2 immune related myocarditis;
9. Patients with active or ever suffered from autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except patients with clinically stable autoimmune thyroid disease and type I diabetes.
10. Have received systemic corticosteroid (prednisone>10mg/day or equivalent doses of similar drugs) or other immunosuppressive therapy within 14 days prior to the first use of the study drug; Excluding the following situations: treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; Short term use of glucocorticoids for preventive treatment (such as preventing contrast agent allergies).
11. History of esophageal and gastric varices, severe ulcers, unhealed wounds, abdominal fistulas, abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to the first administration; History of gastrointestinal perforation and/or fistula, gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), and extensive intestinal resection (partial colectomy or extensive small bowel resection) within 6 months prior to the first administration;
12. Severe infections, including but not limited to bacteremia, severe pneumonia, or other serious infection complications requiring hospitalization, occurred within 4 weeks prior to the start of the study treatment; Within 2 weeks prior to the first administration, there is an active infection with CTCAE ≥ 2 that requires intravenous anti infective treatment;
13. History of immunodeficiency, including HIV testing positive; Presence of active hepatitis B (HBV DNA higher than the upper limit of normal values in the research center) or hepatitis C (anti HCV positive and HCV RNA higher than the lower limit of analysis method detection);
14. Individuals with active pulmonary tuberculosis infection detected through medical history or CT examination within the year prior to enrollment, or those with a history of active pulmonary tuberculosis infection more than one year ago but without formal treatment;
15. Adverse reactions to previous anti-tumor treatments have not yet recovered to a CTCAE v 5.0 rating of ≤ 1 (except for hair loss, grade 2 peripheral neurotoxicity, meeting the numerical requirements of the inclusion criteria, or other situations determined by the researcher to not affect the study drug treatment);
16. Have received chemotherapy within 3 weeks prior to the first use of the investigational drug, and have received large molecule biologic therapy (including immunotherapy) or other non marketed clinical investigational drug therapy or other anti-tumor treatments within 4 weeks prior to the first use of the investigational drug; Excluding the following:

    1. Oral fluorouracil and small molecule targeted drugs should be administered within 2 weeks before the first use of the investigational drug or within 5 half lives of the drug (whichever is longer);
    2. Traditional Chinese medicine with anti-tumor indications should be used 2 weeks before the first use of the investigational drug;
    3. Radical radiotherapy is administered 4 weeks before the first use of the study drug, while palliative radiotherapy is administered 2 weeks before the first use of the study drug; During the efficacy expansion phase, those who have been treated with immune checkpoint agonists (such as CD137 agonists) or immune checkpoint inhibitors (such as PD-1, PD-L1, etc.) within 6 months prior to the first use of the investigational drug are not allowed to be enrolled.

18. Have undergone major organ surgery within 4 weeks prior to the first use of the investigational drug, have experienced significant trauma, or require elective surgery during the trial period; Perform coarse needle aspiration biopsy or other minor surgery within 7 days before the first medication (excluding central venous catheterization and infusion port implantation); 19. Within 4 weeks before the first administration, there is a history of bleeding tendency or coagulation disorders and/or clinically significant bleeding symptoms or risks, including but not limited to: a Gastrointestinal bleeding; b. Hemoptysis (coughing up ≥ 15ml of fresh blood or blood clots); c. Nasal bleeding/epistaxis; d. Receive therapeutic anticoagulant therapy before the first administration; 20. History of hypertensive crisis or hypertensive encephalopathy in the past; Within one month before the first administration, there is hypertension and the systolic blood pressure is ≥ 150mmHg or diastolic blood pressure is ≥ 100mmHg after oral antihypertensive medication; 21. Active or previous history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea); 22. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 23. Known to have a history of severe allergic reactions to multiple medications; 24. Receive live virus vaccine 30 days before the first administration, or plan to receive live vaccine during the study period; According to the researchers' assessment, there are other factors that may affect the research results or force the termination of this study, such as alcohol abuse, drug abuse, other serious illnesses (including mental illnesses) that require concomitant treatment, severe abnormal laboratory test values, family or social factors, and other situations that may affect the safety of the subjects or the collection of experimental data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2028-05-20 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
DLT of CVL006 monotherapy in advanced solid tumor patients. | In Phase Ia trials, if there is a delay in the second administration 28 days after the first dose, the DLT observation period will be extended to 14 days after the second administration.
  Safety events that occur during the DLT observation period and are determined by researchers to be related to the investigational drug.
MTD of CVL006 monotherapy in patients with advanced solid tumors. | Phase Ia trial, from the first subject to the end of the DLT observation period for the last subject.
  During the DLT observation period, the highest dose at which ≤ 1 subject experienced DLT and could not continue to increase in dose among at least 6 subjects
RP2D of CVL006 monotherapy in patients with advanced solid tumors | From the first subject enrolled in Phase 1a to the last subject removed from Phase Ib.
  RP2D is an extended study conducted through dose escalation stage exploration, recommended by SMC, to obtain sufficient safety, tolerability, PK, and preliminary efficacy results. The dosage selected for subsequent efficacy expansion stage is further discussed and confirmed by SMC. RP2D should not exceed the MTD obtained by dose escalation.

SECONDARY OUTCOMES:
Objective response rate (ORR) in patients | Throughout the study for approximately 5 years.
  ORR by investigator
Progression-free survival (PFS) | Throughout the study for approximately 5 years.
  Progression-free survival (PFS), defined as the time from the start of study treatment to any documented tumor progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Throughout the study for approximately 5 years.
  Overall survival (OS), defined as the time from enrollment to death due to any cause. Efficacy of each tumor type will be analyzed independently.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai GoBroad Cancer Hospital China Pharmaceutical University

IPD SHARING:
Plan to Share IPD: No